CLINICAL TRIAL: NCT00657683
Title: A Phase I, Randomized, Single-blind, Controlled, Single Center Study to Evaluate the Safety and Immunogenicity of a Dose Range of a Glycoconjugate Antigen Vaccine of Group B Streptococcus in Healthy Women 18-40 Years of Age
Brief Title: A Phase I, Randomized, Single-blind, Controlled, Single Center Study to Evaluate the Safety and Immunogenicity of a Dose Range of a Monovalent Glycoconjugate Antigen Vaccine of Group B Streptococcus in Healthy Women 18-40 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V98P1
Record Dates: First submitted 2008-03-27; First posted 2008-04-14 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Invasive Group B Streptococcus (GBS) Disease
Keywords: GBS; GBS prevention
MeSH Terms: conditions — Guillain-Barre Syndrome; Disease

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Monovalent GBS-CRM glycoconjugate vaccine
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Monovalent GBS-CRM glycoconjugate vaccine — 1 dose of GBS conjugate vaccine
  Arms: 1
Biological: Placebo — 1 dose of placebo
  Arms: 2

SUMMARY:
The goals of the proposed study are to evaluate the safety, tolerability and immunogenicity of a GBS vaccine. Previous studies suggest that immune responses against GBS can protect humans from infection.

ELIGIBILITY:
Inclusion Criteria:

* healthy females 18 through 40 years of age;
* have provided written informed consent after the nature of the study has been explained;
* are available for all visits scheduled for the study (i.e. are not planning to leave the area before the end of the study period);
* are in good health as determined by: medical history, physical assessment, clinical judgment of the investigator

Exclusion Criteria:

* unwilling or unable to give written informed consent to participate in the study;
* pregnant (serum pregnancy test)
* unwilling to use acceptable birth control from screening and until at least 3 months after the final immunization
* nursing (breastfeeding) mothers

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of an intramuscular GBS conjugate vaccine. Safety will be assessed by measuring the incidence of local and systemic reactogenicity, adverse events and serious adverse events. | 1 month

SECONDARY OUTCOMES:
To study the magnitude and durability of GBS-specific antibody responses over 12 months. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Institute for Pharmacokinetic and Analytical Studies, I.P.A.S. S.A., Ligornetto, Switzerland